CLINICAL TRIAL: NCT05866783
Title: Serum Glycomics as Prognostic and Diagnostic Biomarkers of Disease Recurrence in Liver Transplant Recipients With Hepatocellular Carcinoma
Acronym: GLITCA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Hospital, Antwerp (Other); Universitaire Ziekenhuizen KU Leuven (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0492
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Prognostic Biomarker; Liver Transplantation; Diagnostic Biomarker; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No HCC recurrence: Patients receiving a liver transplantation that do NOT develop HCC recurrence after liver transplantation.
  Interventions: Diagnostic Test: HCCRecurrencePrognosticScore; Diagnostic Test: HCCRecurrenceDiagnosticScore
- HCC recurrence: Patients receiving a liver transplantation that develop HCC recurrence after liver transplantation.
  Interventions: Diagnostic Test: HCCRecurrencePrognosticScore; Diagnostic Test: HCCRecurrenceDiagnosticScore

INTERVENTIONS:
Diagnostic Test: HCCRecurrencePrognosticScore — Determination of serum glycomics pre-transplant using an optimal cutoff based on statistic modeling
Diagnostic Test: HCCRecurrenceDiagnosticScore — Determination of serum glycomics post-transplant using an optimal cutoff based on statistic modeling

SUMMARY:
Liver transplantation (LT) is the only curative option for a selection of patients with hepatocellular carcinoma (HCC) based on clinical selection criteria known as the Milan criteria. Nevertheless, 15% of these patients still show tumour recurrence after LT. In a monocentric pilot study, we have demonstrated that specific changes in N-glycan profiles (measured before LT) occur in HCC patients receiving LT1. These specific changes proved to be strongly associated with the risk of HCC recurrence and overall death after LT, independent of the criteria used for stringent patient selection. Pathophysiologically, it is known that abberations in protein glycosylation are involved in the onset en development of HCC. As such, a prognostic biomarker was developed that can clearly differentiate between patients with and without increased risk of HCC recurrence.

The primary goal of this research study is to set up a prospective, multicentre study in order to validate the prognostic value of this glycomics-based serum biomarker. As such, the risk of tumour recurrence in patients undergoing LT for HCC will be estimated independent from the Milan criteria and the French alpha-fetoprotein model as the current standard. The secondary goal is to explore the potential of serum glycomics as markers of early recurrence after LT for HCC. More specifically, we aim to investigate whether serial glycomics determination at fixed time points after LT could allow early detection of recurrent HCC even before it is visible on conventional imaging. Consequently, a diagnostic biomarker for monitoring early recurrence after LT could be developed with the potential of redirecting treatment strategies already in an early disease stage.

In case the promising data from the pilot study will be confirmed, the prognostic biomarker could be implemented in daily clinical practice leading to optimization of patient selection using a simple blood test before LT. More specifically, this marker could improve organ allocation thus preventing unnessecary treatment toxicity for the patient and reducing the costs of treatment for society. Moreover, it should be emphasized that a patent application was already submitted and accepted in collaboration with TechTranfer of Ghent University (PCT/EP2021/057788-Prognostic markers of disease recurrence in liver transplant recipients with hepatocellular carcinoma).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated patient informed consent document
* Diagnosis of hepatocellular carcinoma
* Age ≥ 18 years
* Ability to comply with protocol-specified evaluations and scheduled visits
* Eligible for liver transplantation and/or active on the waiting list for liver transplantation
* Consulted the department of Gastroenterology and Hepatology

Exclusion Criteria:

* Diagnosis of other liver tumors (eg. liver metastasis, cholangiocarcinoma)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with hepatocellular carcinoma active on the waiting list or undergoing a liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2038-01-01 (Estimated)

PRIMARY OUTCOMES:
HCC recurrence | 18 months
Disease-free survival | 18 months

SECONDARY OUTCOMES:
Overall survival | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided